CLINICAL TRIAL: NCT00812227
Title: Neural Correlates of Psychodynamic Psychotherapy for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Hope for Depression Research Foundation (Other)
Responsible Party: Principal Investigator, Joshua L. Roffman MD, MMSc, Staff psychiatrist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-P-001181
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Psychotherapy; Neuroimaging; Subjects with Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Psychotherapy, Psychodynamic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psychodynamic psychotherapy (Experimental)
  Interventions: Behavioral: Psychodynamic Psychotherapy

INTERVENTIONS:
Behavioral: Psychodynamic Psychotherapy — Screened and eligible patients will receive 16 individual sessions of psychodynamic psychotherapy, each lasting 45-50 minutes.

SUMMARY:
The purpose of this study is to see whether we can predict which patients with depression will get better when we treat them with psychodynamic psychotherapy. We will use neuroimaging (a method of looking at brain activity) in this study. We want to see whether there are changes in the brains of patients receiving this type of therapy. We hypothesize that these changes may predict how well certain parts of the psychotherapy treatment process works.

DETAILED DESCRIPTION:
In this study, we will treat patients with brief psychodynamic psychotherapy. Psychodynamic psychotherapy is a type of treatment that may be as helpful as medications in treating depression. It focuses on thoughts, feelings, and behaviors as well as both current and past relationships. Psychotherapy explores better ways of coping with feelings, expressing needs, and interacting with others in order to cope with depression and other life problems. Subjects will go to 16 weekly, 45-minute, individual sessions of psychodynamic psychotherapy over the course of the study. At five times throughout the study, subjects will come in for extra visits, which last approximately 1.5 hours and which include: speaking with a study doctor about depressive symptoms, filling out extra questionnaires, and performing positron emission tomography (PET)and a Quantitative Electroencephalogram (QEEG). The QEEG is a machine that measures the electrical activity of the brain. This task will take approximately 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be adults, ages 18 to 60 years;
* Able to provide written informed consent;
* MDD, current according to the fourth version of the Diagnostic and Statistical Manual for Mental Disorders (DSM-IV);
* QIDS-SR score of >= 12 at screen;
* Current major depressive episode (MDE) length of < 5 year;
* Treated with an SSRI, SNRI, or bupropion at adequate doses (defined as 20 mg/day or more of fluoxetine, citalopram, or paroxetine; 10 mg/day or more of escitalopram; 50 mg/day or more of sertraline; 75 mg/day or more of venlafaxine; 15 mg/day of mirtazapine; or 40 mg/day of duloxetine; or 100mg/day of bupropion(wellbutrin)) during the current episode for at least 8 weeks; and,
* At the time of screen visit, patients must be on a stable dose of SSRI, SNRI, or bupropion for the past 4 weeks.

Exclusion Criteria:

* Pregnant women or women of child bearing potential who are not using a medically accepted means of contraception (to include oral contraceptive or implant, condom, diaphragm, spermicide, intrauterine device, tubal ligation, or a partner with vasectomy). Women of childbearing age who wish to enter the study will be required to undergo a pregnancy test (beta-HCG) prior to initiating treatment; an additional blood pregnancy test (beta HCG) will be completed if subject wants to do PET scan
* Patients who, in the investigator's judgment, pose a current, serious suicidal or homicidal risk. These patients will be immediately referred to appropriate clinical treatment;
* Patients who, in the opinion of the therapist, are not depressed at the time of their first psychotherapy visit;
* Patients who are currently being treated by a psychotherapist individually or who have received individual psychotherapy during the past 6 months. Couples therapy and family therapy will not be considered exclusionary criteria;
* Patients with neurological illnesses, including a history of seizure or head trauma with loss of consciousness;
* Patients with unstable diabetes, kidney disease, or significant medical illness;
* Patients with history of allergy to FDG
* The following DSM-IV diagnoses: substance use disorders active within the last six months, any bipolar disorder (current or past), any psychotic disorder (current or past), any post-traumatic stress disorder (current or past), any obsessive compulsive disorder (current or past), or any panic disorder (current, past allowed). Generalized anxiety disorder or adjustment disorder are not exclusionary;
* Patients currently requiring other psychotropic medications, including anticonvulsants, benzodiazepines, antipsychotics, stimulants, or sedative hypnotics (other than diphenhydramine);however, patients will be permitted to take trazodone in addition to their primary antidepressant if it is taken as a sleep aid, rather than a primary antidepressant;
* Psychotic features in the current episode, or a history of psychotic features, as assessed by SCID;
* Patients who have undergone > 3 previous adequate attempts at psychodynamic psychotherapy (deemed "adequate" by the screening physician), which were considered unhelpful or unsuccessful by patient report (according to patient report);
* Patients with a history of antidepressant-induced hypomania; and
* Patients with a history of medication non-compliance.
* Patients with Axis II pathology (personality disorder) that, in the opinion of the screening physician, would interfere with subjects' ability to participate in the treatment and/or comply with the protocol, such as severe borderline or narcissistic personality disorder.
* Patients who have had electroconvulsive therapy (ECT) within the 12 months preceding baseline

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2008-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Correlation between changes in HAMD-17 and changes in QEEG measurements (theta cordance) from treatment initiation to two weeks after starting treatment | Weeks 0 through 16
PET: Treatment-related change in FDG metabolism within regions-of-interest identified at baseline as related to depression severity. | Week 0, Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Roffman, MD, Principal Investigator — Massachusetts General Hospital Department of Psychiatry; Janet Witte, MD, MPH, Principal Investigator — Massachusetts General Hospital Department of Psychiatry
Locations (1):
- Depression Clinical and Research Program, Boston, Massachusetts, United States